CLINICAL TRIAL: NCT04348240
Title: Transmissibility and Viral Load of SARS-CoV-2 Through Oral Secretions
Brief Title: Transmissibility and Viral Load of SARS-CoV-2 in Oral Secretions
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200094; 20-D-0094
Record Dates: First submitted 2020-04-15; First posted 2020-04-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: COVID-19
Keywords: Saliva; Coronavirus; SARS-CoV-2; Symptoms; COVID19; Natural History
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: asymptomatic or mildly symptomatic high-risk subjects with unknown SARS-CoV-2 status but with known history of close personal contact with a COVID-19 positive person.
- Group 2: asymptomatic or mildly symptomatic (e.g., low grade fever, mild malaise, minor sore throat, runny nose, or sneezing) subjects who are COVID-19 positive.
- Group 3: COVID-19 positive individuals retesting negative can be enrolled to complete the electronic questionnaire(s) and allow evaluation of history of symptoms.
- Group 4: COVID-19 positive individuals enrolled and admitted to the NIH Clinical Center for other protocols.

SUMMARY:
Background:

COVID-19 is a worldwide pandemic and currently there is no effective therapy or vaccine. SARS-CoV-2, the virus that causes the COVID-19 respiratory infection, appears to be very contagious however all the modes of transmission are unclear. Transmission may occur in up to 25 percent of cases when there are no symptoms (asymptomatic). Before there are any symptoms, droplet spray during speaking may increase transmission from person to person; most of the spray is saliva. Researchers at the NIH would like to test saliva for the virus before symptoms are reported. Additionally, they would like to examine the importance of using masks to prevent transmission. They hope to better understand how COVID-19 is spread among people and how it can be prevented. For this study they would like to collect samples from the nose (nasopharyngeal swab), mouth (spit sample), eye (conjunctival fluid) and blood to test for the virus and if it is contagious.

Objectives:

To determine if the SARS-CoV-2 virus is present in saliva in asymptomatic individuals who are COVID-19 positive. To determine if using masks can prevent transmission.

Eligibility:

People ages 18 and older without symptoms or with mild symptoms (e.g., low grade fever,

mild malaise, minor sore throat, runny nose, or sneezing) who have been in close contact (e.g. live in the same house) with someone who has tested positive for COVID-19 or people who have tested positive for COVID-19 and have mild (e.g., low grade fever, mild malaise, minor sore throat, runny nose, or sneezing) or no symptoms.

Design and Procedures:

For screening, interested participants will contact a study team member. The interested participant will be asked to provide documentation of COVID-19 positive status, their symptoms, or their contact to a COVID-19 positive person.

Participants will be asked to come to the NIH drive-up COVID-19 testing site or NIH Clinical Center (Bethesda, MD) for 2 or more visits in 15 days for the following procedures: nasal swab for COVID-19 and viral load, verbal symptom assessment, saliva collection, and speaking exercise to capture oral fluid. During this time, participants will also be asked to participate in phone calls with the study staff and to complete questionnaires electronically. Participants will have weekly telephone calls to discuss their symptoms and 2-5 drive-up visits to the NIH within 28 days. If visits are scheduled at the Clinical Center, participants will have the option to participate in providing blood sample(s), a conjunctival swab and 1-2 salivary gland biopsies.

If a participant has tested positive, they may be asked to return to the NIH after they have recovered from COVID-19 for additional sampling.

The following procedures are part of this research:

* Speaking exercise - participants will be asked to read a short script with and without wearing a mask. The droplets they produce while they speak will be collected.
* Saliva collection - participants will spit into a cup and have saliva collected from different areas of the mouth. They should not eat 90 minutes before this but drinking water or juice is acceptable. They may have their tongue painted with a sour liquid to increase their saliva.
* Nasal swab- participants will have a swab rubbed inside their nose.
* Nasopharyngeal swab - participants that are close contacts of COVID-19 positive individual(s) and need a COVID-19 test, will have a swab inserted through the nose to rub the back of their throat.
* Questionnaires - participants will complete questionnaires about their symptoms electronically at home.

The following procedures are optional for participants to agree to participate in and will be performed in the Clinical Center:

* Blood sample(s) - participants will have blood collection via venipuncture.
* Conjunctival swab - participants will have the inner lower eyelid wiped with swab.
* Minor salivary gland biopsy - participants will have tiny glands in mouth removed. Procedure will be done in the hospital.

Participants will be paid up to a total of $300 for the study, based on the number of visits to NIH and the types of procedures performed. Payment will be: $50 on Day 1, Day 15 and at the recovery visit. Participants who agree to the optional conjunctival swab and/or biopsy will be paid $50 for each conjunctival swab (up to 1) and/or $50 for each salivary biopsy (up to 2).

If at any time the participants start to have moderate or severe respiratory symptoms, their participation in the study will end and they should seek care with their local provider.

DETAILED DESCRIPTION:
COVID-19 is a worldwide pandemic without an effective therapy. A series of reports have implicated that asymptomatic transmission occurs in at least 25% SARS-CoV-2 cases. We hypothesize that droplet emission from oral fluids generated during speaking could be an important and actionable factor driving asymptomatic transmission. We aim to collect oral and nasal secretions, conjunctival fluid and blood to test for viral load and viral infectivity in 1) asymptomatic or mildly symptomatic high-risk subjects with unknown SARS-CoV-2 status, but with a history of close personal contact with a SARS-CoV-2 positive person and 2) asymptomatic or mildly symptomatic subjects who are SARS-CoV-2 positive. 3) COVID-19 positive individuals retesting as negative can be enrolled to complete the electronic questionnaire(s) assessment and allow for evaluation of history of symptoms. 4) COVID-19 positive individuals admitted to the NIH Clinical Center can be enrolled as a symptomatic comparison cohort.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all the following criteria:

1. Willing and able to sign and date the informed consent form
2. Willing to comply with all study procedures and available for study visits and calls
3. Male or female, aged >= 18 years of age
4. Persons who test COVID-19 positive in past 48 hours (verbal confirmation followed by documented test results, sent electronically) and are asymptomatic or have mild symptoms (e.g., fever, mild malaise, sore throat or sneezing) individuals who have re-tested and are negative may be enrolled to understand progression and resolution of disease; persons hospitalized at the NIH Clinical Center meeting Inclusion Criteria 1-3 may be enrolled on this study
5. Persons considered high risk for COVID-19 due to personal contact within the past 7 days with a COVID-19 positive individual (e.g., co-habitating family member of COVID-19 positive) and has no symptoms or mild symptoms of COVID-19 - verbal confirmation followed by documented test results of positive individual, sent electronically

EXCLUSION CRITERION:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. COVID-19 positive subjects with active moderate or severe symptoms of cough or shortness of breath (upper and lower respiratory symptoms) or currently requiring hospitalization at a hospital other than NIH Clinical Center (recovering COVID-19 positive patients can be enrolled).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1) asymptomatic high-risk subjects with known history of close personal contact with a COVID-19 positive person not tested (SARS-CoV2 status unknown)2) asymptomatic or mildly symptomatic (fever withoutcough, sneezing or shortness of breath) subjects who are COVID-19 positive 3) COVID-19 positive individuals retesting negative can be enrolled to complete the electronic questionnaire(s) assessment and allow evaluation of history of symptoms. 4) COVID-19 positive individuals enrolled and admitted to the NIH Clinical Center for other protocols.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
To determine SARS-CoV-2 viral load and infectivity insaliva that may contribute to asymptomatic transmission
  detection of virus in saliva, blood and conjunctival fluid

CONTACTS AND LOCATIONS:
Overall Officials: Blake M Warner, D.D.S., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Rubin EJ, Baden LR, Morrissey S. Audio Interview: Lessons from Covid-19 Hotspots. N Engl J Med. 2020 Apr 2;382(14):e35. doi: 10.1056/NEJMe2007783. No abstract available. PMID 32242382
- [Background] Fauci AS, Lane HC, Redfield RR. Covid-19 - Navigating the Uncharted. N Engl J Med. 2020 Mar 26;382(13):1268-1269. doi: 10.1056/NEJMe2002387. Epub 2020 Feb 28. No abstract available. PMID 32109011
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-D-0094.html